CLINICAL TRIAL: NCT07027306
Title: The Osteoporotic Fracture Classification-based Scoring System for Treatment Decision in Thoracolumbar Osteoporotic Fractures: An International Multicenter Prospective Study
Brief Title: The Osteoporotic Fracture Classification-based Scoring System for Treatment Decision in Thoracolumbar Osteoporotic Fractures
Status: Not yet recruiting | Type: Observational
Sponsor: AO Foundation, AO Spine (Other)
Responsible Party: Sponsor
Other Study IDs: TL-OF
Record Dates: First submitted 2025-05-02; First posted 2025-06-18 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Osteoporotic Fractures; Osteoporosis
MeSH Terms: conditions — Osteoporotic Fractures; Osteoporosis | interventions — Pedicle Screws; Kyphoplasty; Vertebroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OF score accordance group: Initial treatment decision in accordance with the OF score recommendations
  Interventions: Procedure: Posterior stabilization (pedicle screws)
- OF score discordance group: Initial treatment decision in discordance with the OF score recommendations
  Interventions: Procedure: Posterior stabilization (pedicle screws)

INTERVENTIONS:
Procedure: Posterior stabilization (pedicle screws) — * Any other type of solely vertebral augmentation (stents, etc.), specify
  * Posterior stabilization (pedicle screws)
  * Posterior stabilization (pedicle screws) with kyphoplasty/vertebroplasty
  * Posterior stabilization (pedicle screws) with screw augmentation
  * Posterior stabilization (pedicle screws) with screw augmentation and kyphoplasty/vertebroplasty
  * Posterior stabilization (pedicle screws) with vertebral osteotomy (pedicle subtraction osteotomy or similar)
  * Combined posterior and anterior stabilization
  Other Names: Kyphoplasty; Vertebroplasty

SUMMARY:
This is an international multicenter prospective observational study. Patients with radiologically confirmed, symptomatic, single- or multilevel contiguous TL (from T1 to L5) fractures as a result of primary osteoporosis will be recruited from participating clinics/hospitals (ie, study sites). Fractures included are insufficiency fractures (confirmed by magnetic resonance imaging [MRI]) and traumatic fractures (low-energy trauma, confirmed by computed tomography [CT] or MRI).

DETAILED DESCRIPTION:
This is an international multicenter prospective observational study. Postmenopausal women ≥ 50 years old and men > 60 years old with radiologically confirmed, symptomatic, single- or multilevel contiguous TL (from T1 to L5) fractures as a result of primary osteoporosis will be recruited from participating clinics/hospitals (ie, study sites). Fractures included are insufficiency fractures (confirmed by magnetic resonance imaging [MRI]) and traumatic fractures (low-energy trauma, confirmed by computed tomography [CT] or MRI).

All osteoporotic TL fractures will be classified using the OF classification system (OF 1 to OF 5). Only the most severe fracture will be used to calculate the OF score. The OF score will be subsequently calculated to aid the surgeons' decision making on the initial treatment plan, which is categorized as either nonsurgical or surgical treatment.

To address the primary study objective, depending on whether the treating surgeons' eventual initial treatment decisions agree with the OF score recommendations, patients will be divided into two groups: 1) patients whose initial treatment is in accordance with the OF score recommendations (the Accordance group), and 2) patients whose initial treatment is in discordance with the OF score recommendations (the Discordance group). Accordance refers to 1) when the OF score is > 6, surgical treatment is prescribed by the treating surgeons, 2) when the OF score is < 6, nonsurgical treatment only is prescribed by the treating surgeons, and 3) when the OF score is 6, either surgical or nonsurgical treatment is prescribed (Note: any surgeons' decision is deemed in accordance with the OF score as the system leaves the decision to the surgeons' discretion in this situation).

Accordance/Discordance group assignment is based on the agreement/discrepancy between the eventual treatment and the recommendations from the OF score that is obtained up to Day 0, although OF scores may be calculated at follow-ups (FUs) for subsequent treatment decision making (eg, whether the treatment plan needs to be modified).

Depending on the actual initial treatment assigned to the patients by the treating surgeons, patients will be divided into two groups: 1) patients assigned to receive nonsurgical treatment (the Nonsurgical group), and 2) patients assigned to receive surgery (the Surgical group).

Day 0 refers to the day when the initial treatment is decided and starts (categorized as nonsurgical or surgical treatment). Subsequent FUs will be calculated in reference to Day 0. Patients will be followed up clinically at discharge, 6 weeks, 3 months, 6 months, and 12 months.

The primary outcome of the study is the return to the mobility level before the injury or symptom onset (as reported by the patient). The FU period for the primary endpoint of the study is 3 months (short-term), and 12 months for the secondary endpoints (long-term).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women ≥ 50 years old or men > 60 years old

  o Menopause refers to amenorrhea for 1 complete year.
* Radiologically confirmed new diagnosis of symptomatic, single or multilevel TL (from T1 to L5) fractures, ie, the index fracture(s).

  * In case of a multilevel fracture, the fracture must be contiguous.
  * The index fracture is confirmed by MRI as an insufficiency (or fragility) fracture or is confirmed by CT or MRI as traumatic fracture (low-energy trauma)
* The index fracture(s) is a result of primary osteoporosis. Diagnosis of primary osteoporosis is based on any of the followings in the absence of causes for secondary osteoporosis (such as long-term use of steroids, rheumatoid arthritis, type 1 diabetes mellitus [DM], and other metabolic bone disorders [eg, rickets/osteomalacia, Paget's disease, osteogenesis imperfecta, and primary hyperparathyroidism]) [13-15]:

  * A T-score ≤ -2.5 in the lumbar spine, femoral neck, total hip, or 1/3 radius
  * Presence of fragility fracture (either a previous fragility fracture or the index fracture is a fragility fracture). Fragility fractures are fractures due to no or low-energy trauma, eg, slips, trips, or falls from less than double the body height, and heavy lifting.
* The index osteoporotic TL fracture being classified based on the OF Classification from OF 1 to OF 5:

  * OF 1: No deformation (vertebral body edema on MRI using short tau inversion recovery [STIR] sequence)
  * OF 2: Deformation of one endplate
  * OF 3: Deformation of one endplate with distinct posterior wall involvement
  * OF 4: Deformation of both endplates with/without posterior wall involvement
  * OF 5: Injuries with anterior or posterior tension band failure
* Ability to provide informed consent according to the EC/IRB defined and approved procedures

Exclusion Criteria:

* Patients with spinal tumors
* Patients with concomitant cervical fractures
* Patients showing any signs of spinal infections
* Patients with fractures due to high-energy or high-impact trauma, eg, a fall from double the body height or higher, motor vehicle accident with > 100 km/h in cars with airbags, or motor vehicle accident > 50 km/h without airbags, polytrauma
* Patients with concomitant fracture in the pelvis, upper extremities, and/or lower extremities which could affect the main study outcomes (specifically, patient mobility and pain)
* Patients for whom no FUs are possible
* Previous instrumented surgery in the affected spine levels
* Patients with single-level fracture or contiguous multilevel fracture adjacent to previous instrumented surgery
* Patients who are mentally impaired and therefore not able to adhere to the study procedures and data collection
* Patients who are bedridden before the index fracture
* Recent history of substance abuse (ie, recreational drugs and alcohol) that would preclude reliable assessments
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women ≥ 50 years old or men > 60 years old
Sampling Method: Non-Probability Sample
Enrollment: 648 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Return to mobility | 3 moths post-operative
  Determination in patients with symptomatic osteoporotic TL fractures whether an initial treatment adhering to the OF score recommendations (the Accordance group) generates better short-term patient outcomes regarding time to return to mobility level before injury or symptom onset within 3 months after treatment compared to an initial treatment decision not adhering to the OF score recommendations (the Discordance group).
  The primary outcome of the study is return to the mobility level. Patients will be instructed to evaluate their overall mobility level in reference to their pre-injury or pre-symptom mobility status. This primary outcome will be reported by the patient and measured on a continuous scale of 0 to 100 (0 = no return at all, 100 = full return).
  Primary endpoint of the study is the time (days) to return of pre-injury or pre-symptom mobility level within 3 months after Day 0. Threshold of returning is defined as ≥ 80 on the continuous scale.

SECONDARY OUTCOMES:
Comparison of return to mobility (categorical scale) | 3 months post-operative and 12-months postoperative
  To compare the proportion (in percentage) of patients returning to mobility level (measured in 4 categories: Not at all returned, Partially returned with major restrictions, Partially returned with minor restrictions, and Fully returned) at 3 months (short-term outcome) and 12 months (long-term outcome) between the Accordance and the Discordance group.
Comparison of the extent of return to mobility | 3 months post-operative and 12-months postoperative
  To compare the extend of return (measured on a continuous scale of 0 to 100, with 0 representing no return at all and 100 representing full return) at 3 months (short-term outcome) and 12 months (long-term outcome) between the Accordance and the Discordance group.
Comparison of clinical outcome | 3 months post-operative and 12-months postoperative
  To compare the clinical outcome at 3 and 12 months between the Accordance and the Discordance groups, between patients whose initial and subsequent treatment decisions adhere to the OF score recommendations and those whose treatment decisions do not completely adhere to the OF score recommendations, between patients with symptomatic osteoporotic TL fracture treated non-surgically and those treated surgically and between nonsurgical and surgical treatments (as determined by a blinded expert group). Clinical outcome defined as any of the following events occurring: New or adjacent vertebral fracture, crossover to surgery or additional surgery, use of analgesic, fracture- or treatment-related adverse events.
Comparison of the proportion return to mobility | 3 months post-operative and 12-months postoperative
  To compare the proportion of patients returning to pre-injury mobility level at 3 and 12 months between the Accordance and the Discordance groups, between patients whose initial and subsequent treatment decisions adhere to the OF score recommendations and those whose treatment decisions do not completely adhere to the OF score recommendations, between patients with symptomatic osteoporotic TL fracture treated non-surgically and those treated surgically and between nonsurgical and surgical treatments (as determined by a blinded expert group).
Comparison of Timed Up & Go test | 3 months post-operative and 12-months postoperative
  To compare timed Up & Go in seconds at 3 and 12 months between the Accordance and the Discordance groups, between patients whose initial and subsequent treatment decisions adhere to the OF score recommendations and those whose treatment decisions do not completely adhere to the OF score recommendations, between patients with symptomatic osteoporotic TL fracture treated non-surgically and those treated surgically and between nonsurgical and surgical treatments (as determined by a blinded expert group).
Comparison of daily activities | 3 months post-operative and 12-months postoperative
  To compare the score of the Barthel Index (ranging from 0 to 100, with higher scores indicating greater functional independence) at 3 and 12 months between the Accordance and the Discordance groups, between patients whose initial and subsequent treatment decisions adhere to the OF score recommendations and those whose treatment decisions do not completely adhere to the OF score recommendations, between patients with symptomatic osteoporotic TL fracture treated non-surgically and those treated surgically and between nonsurgical and surgical treatments (as determined by a blinded expert group).
Comparison of pain NRS (Numeric Rate Scale) | 3 months post-operative and 12-months postoperative
  To compare the score of pain Numeric Rate Scale (ranging from 0 to 10, with 0 representing no pain and 10 the worst imaginable pain) at 3 and 12 months between the Accordance and the Discordance groups, between patients whose initial and subsequent treatment decisions adhere to the OF score recommendations and those whose treatment decisions do not completely adhere to the OF score recommendations, between patients with symptomatic osteoporotic TL fracture treated non-surgically and those treated surgically and between nonsurgical and surgical treatments (as determined by a blinded expert group).
Comparison of ODI (Oswestry Disability Index) | 3 months post-operative and 12-months postoperative
  To compare the score of ODI (ranging from 0 to 100%, with higher scores indicating greater disability) at 3 and 12 months between the Accordance and the Discordance groups, between patients whose initial and subsequent treatment decisions adhere to the OF score recommendations and those whose treatment decisions do not completely adhere to the OF score recommendations, between patients with symptomatic osteoporotic TL fracture treated non-surgically and those treated surgically and between nonsurgical and surgical treatments (as determined by a blinded expert group).
Comparison of quality of live | 3 months post-operative and 12-months postoperative
  To compare the score of EQ-5D-5L (ranging from 0 to 1, with 0 representing death and 1 perfect health) at 3 and 12 months between the Accordance and the Discordance groups, between patients whose initial and subsequent treatment decisions adhere to the OF score recommendations and those whose treatment decisions do not completely adhere to the OF score recommendations, between patients with symptomatic osteoporotic TL fracture treated non-surgically and those treated surgically and between nonsurgical and surgical treatments (as determined by a blinded expert group).
Comparison of the AO Spine PROST | 3 months post-operative and 12-months postoperative
  To compare the score of AO Spine PROST (ranging from 0 to 100, with higher score indicating better recovery of functional level before trauma) at 3 and 12 months between the Accordance and the Discordance groups, between patients whose initial and subsequent treatment decisions adhere to the OF score recommendations and those whose treatment decisions do not completely adhere to the OF score recommendations, between patients with symptomatic osteoporotic TL fracture treated non-surgically and those treated surgically and between nonsurgical and surgical treatments (as determined by a blinded expert group).
Comparison of the overall satisfaction | 3 months post-operative and 12-months postoperative
  To compare the proportion of overall satisfaction (measured on a 7-point Likert scale (Extremely satisfied, Very satisfied, Somewhat satisfied, Mixed, Somewhat dissatisfied, Very dissatisfied, Extremely dissatisfied) of patients at 3 and 12 months between the Accordance and the Discordance groups, between patients whose initial and subsequent treatment decisions adhere to the OF score recommendations and those whose treatment decisions do not completely adhere to the OF score recommendations, between patients with symptomatic osteoporotic TL fracture treated non-surgically and those treated surgically and between nonsurgical and surgical treatments (as determined by a blinded expert group).
Complications-determination in relation to surgery | 1 year post-operative
  To determine the rate and type of complications in relation to the type of surgery performed
Complications-determination in relation to OF subtype | 1 year post-operative
  To determine the rate and type of complications in relation to the OF subtype
Determination of type of treatment | 1 year post-operative
  To determine the type of treatment in relation to the OF subtype
Determination of rate and type of surgical treatment | 1 year post-operative
  To determine the type of surgical treatment in relation to the OF subtype. The surgery types are:
  * Kyphoplasty
  * Vertebroplasty
  * Any other type of solely vertebral augmentation (stents, etc.), specify
  * Posterior stabilization (pedicle screws)
  * Posterior stabilization (pedicle screws) with kyphoplasty/vertebroplasty
  * Posterior stabilization (pedicle screws) with screw augmentation
  * Posterior stabilization (pedicle screws) with screw augmentation and kyphoplasty/vertebroplasty
  * Posterior stabilization (pedicle screws) with vertebral osteotomy (pedicle subtraction osteotomy or similar)
  * Combined posterior and anterior stabilization, if yes:
  * Open surgery
  * Percutaneous/minimal-invasive surgery
  * Delete "rate" from 10 only keeping type and list them from above
Proportion between surgery after initial non-surgery treatment | 1 year post-operative
  To determine the proportion of patients who underwent surgery after initial nonsurgical treatment (crossover to surgery).
Agreement between OF classification and investigators | 1 year post-operative
  To determine the proportion of agreement in the OF classification (from OF 1 to OF 5 categories) made by the site investigators and a blinded expert panel.
  OF 1: No deformation (vertebral body edema in MRI-STIR) OF 2: Deformation of one endplate without or with only minor posterior wall involvement OF 3: Deformation of one endplate with distinct posterior wall involvement OF 4: Deformation of both endplates with or without posterior wall involvement OF 5: Injuries with anterior or posterior tension band failure
Validation of AO PROST | 1 year post-operative
  To validate the AO Spine Patient-Reported Outcome Spine Trauma (PROST) in terms of interpretability, internal consistency, and responsiveness in patients with symptomatic osteoporotic TL fractures.
  The AO Spine PROST consists of 19 questions on broad aspects of functioning. Each item has a 0-100 scale, with 0 indicating no function at all and 100 the functional level before trauma. Total score ranges from 0 to 100, with higher score indicating better recovery of functional level before trauma.
Health economic analyses | 1 year post-operative
  To perform health economic analyses to investigate the cost-effectiveness/cost-utility of a) comparing non-surgical to surgical treatment and b) the effect of adhering to the OF score for treating patients with osteoporotic TL fractures compared with not adhering to the OF score.
  The cost-effectiveness will be evaluated using the incremental cost effectiveness ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schnake, MD, Principal Investigator — Center for Spinal and Scoliosis Surgery
Locations (15):
- United States (2):
  - University of California San Francisco (USCF) Department of Orthopaedic Surgery, San Francisco, California
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
- Sanatorio Güemes, Buenos Aires, Argentina
- Cajuru University Hospital, Curitiba, Brazil
- Department of Orthopedic Surgery, Clinica Alemana de Santiago, Santiago, Chile
- Orthopaedic Department, Assiut University Hospitals, Faculty of Medicine, Asyut, Egypt
- Tampere University Hospital, Tampere, Finland
- Center for Spinal and Scoliosis Surgery, Malteser Waldkrankenhaus St. Marien, Erlangen, Germany
- PGIMER - Postgraduate Institute of Medical Education and Research, Chandigarh, India
- Dokkyo Medical University Hospital, Tochigi, Japan
- Island Hospital Spine Centre, George Town, Malaysia
- Spiatlul Clinic De Urgenta, "Profesor Doctor Nicolae Oblu", Iași, Romania
- Security Force Hospital, Riyāḑ, Saudi Arabia
- Spital Emmental - Orthopädie Sonnenhof, Burgdorf, Switzerland
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided